CLINICAL TRIAL: NCT04721691
Title: Efficacy of Epidiolex in Patients With Electrical Status Epilepticus of Sleep (ESES).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Sanjeev Vithal Kothare, Director, Service Line Chief of Child Neurology, Northwell Health
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20-0168
Record Dates: First submitted 2020-09-24; First posted 2021-01-25 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Electrical Status Epilepticus of Slow-Wave Sleep
Keywords: Neurology; Pediatric; ESES
MeSH Terms: interventions — Cannabidiol; Solutions

STUDY DESIGN:
Intervention Model Description: This study aims to assess the efficacy of Epidiolex in patients with ESES. ESES is characterized by sleep potentiated spikes with a spike index greater than 85% (conventional definition) and 50% (new definition). Several drugs including: steroids, intravenous Gama globulin, Clobazam, other benzodiazepines, Valproic acid, and other anti-epileptic drugs have been tried with mixed benefits. Cannabidiol (CBD) would provide a novel mechanism of action to assess for its efficacy in this population4. This will be a double-blind placebo-controlled crossover clinical trial.
Who Masked: Participant, Investigator
Masking Description: All study personnel aside from the institution's pharmacist will remain blinded for the duration of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IP (Active Comparator): Epidiolex (Cannabidiol) is a colorless to yellow solution in a 100mL vial that is to be administered with a 5mL syringe.The starting dosage is 2.5 mg/kg twice daily, or 5 mg/kg/day. After one week, the dosage can be increased to a maintenance dosage of 5mg/kg twice daily, or 10 mg/kg/day. Patients who are tolerating Epidiolex at 10mg/kg per day and require further reduction of seizures may benefit from a dosage increase up to a maximum recommended maintenance. Dosage of 10mg/kg twice daily (20mg/kg/day), in weekly increments of 2.5 mg/kg twice daily(5mg/kg/day), as tolerated. For patients in whom a more rapid titration from 10 mg/kg/day to 20 mg/kg/day is warranted, the dosage may be increased to no more frequently than every other day administration of the 20 mg/kg/day. Dosage resulted in somewhat greater reductions in seizure rates than the recommended maintenance dosage of 10 mg/kg/day, but with an increase in adverse reactions.
  Interventions: Drug: Epidiolex 100 mg/mL Oral Solution
- Placebo (Placebo Comparator): Placebo is a colorless to yellow solution in a 100mL vial that is to be administered with a 5mL syringe. The starting dosage is 2.5 mg/kg twice daily, or 5 mg/kg/day. After one week, the dosage can be increased to a maintenance dosage of 5mg/kg twice daily, or 10 mg/kg/day. Patients who are tolerating Placebo at 10mg/kg per day and require further reduction of seizures may benefit from a dosage increase up to a maximum recommended maintenance. Dosage of 10mg/kg twice daily (20mg/kg/day), in weekly increments of 2.5 mg/kg twice daily(5mg/kg/day), as tolerated. For patients in whom a more rapid titration from 10 mg/kg/day to 20 mg/kg/day is warranted, the dosage may be increased to no more frequently than every other day administration of the 20 mg/kg/day. Dosage resulted in somewhat greater reductions in seizure rates than the recommended maintenance dosage of 10 mg/kg/day, but with an increase in adverse reactions.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Epidiolex 100 mg/mL Oral Solution — Epidiolex is a schedule 5 controlled substance that is a colorless to yellow oral liquid solution that is prepackaged into 100mL vials with 5mL syringes for use. It is typically used for the treatment of seizures associated with Lennox-Gastaut syndrome (LGS) or Dravet Syndrome in patients 2 years of age and older.
  Arms: IP
Other: Placebo — Placebo is composed of dehydrated alcohol, sesame seed oil, strawberry flavor, and sucralose.
  Arms: Placebo

SUMMARY:
This study aims to assess the efficacy of Epidiolex in patients with ESES. ESES is characterized by sleep potentiated spikes with a spike index greater than 85% (conventional definition) and 50% (new definition)1. Several drugs including: steroids, intravenous Gama globulin, Clobazam, other benzodiazepines, Valproic acid, and other anti-epileptic drugs have been tried with mixed benefits2,3. Cannabidiol (CBD) would provide a novel mechanism of action to assess for its efficacy in this population. This will be a double-blind placebo-controlled crossover clinical trial.

DETAILED DESCRIPTION:
This study attempts to view the effect of Epidiolex on subjects with Electrical Status Epilepticus of Sleep (ESES). ESES can cause various types of seizures which can fluctuate during sleep. Similar studies have been conducted with Epidiolex with other seizure disorders such as Lennox-Gastaut syndrome (LGS) and Dravet Syndrome. Since there is no data available on the effect of Cannabidiol (CBD) on patients with ESES, this study hopes to fill that void. As such, patients that have been diagnosed with ESES will be eligible to participate in this study to ascertain whether or not Epidiolex can reduce the frequency or intensity of the seizures brought on by ESES during sleep.

ELIGIBILITY:
In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 2-17 years old
4. In good general health as evidenced by medical history or diagnosed with ESES. "Good health" in relation to this study is understood as stable without current seizures requiring immediate hospitalization.
5. Ability to take oral medication and be willing to adhere to the Epidiolex/Placebo regimen
6. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 1 month after the end of oral Epidiolex administration
7. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner

Exclusion Criteria:An individual who meets any of the following criteria will be excluded from participation in this study:

1. Previous use of cannabidiol within 4 months.
2. Pregnancy or lactation
3. Known allergic reactions to components of the Epidiolex: cannabidiol, sesame seed oil, and sucralose
4. Febrile illness within 1 month of screening
5. Treatment with another investigational drug or other intervention within 6 months
6. Current smoker or tobacco use within 6 months

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Frequency of Spike Wave Index | Up to 20 weeks
  Assess the reduction in spike wave index by evaluating the differences in activity from the four 24-hour ambulatory EEGs each participant obtains while enrolled in this study

SECONDARY OUTCOMES:
Likert Scale Assessment | Up to 20 weeks
  The secondary objective is to assess seizure counts and subjective behavior change on a 5 point Likert scale (1= no improvement, 2= some improvement, 3=moderate improvement, 4=significant improvement, 5=extreme improvement).

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell Health, Lake Success, New York, United States